CLINICAL TRIAL: NCT00165555
Title: Pleurectomy/Decortication Followed by Intrathoracic/Intraperitoneal Heated Cisplatin and Intravenous Sodium Thiosulfate in the Multimodality Treatment of Malignant Pleural Mesothelioma
Brief Title: Pleurectomy/Decortication Followed by Intrathoracic/Intraperitoneal Heated Cisplatin for Malignant Pleural Mesothelioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 99-124
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-03

CONDITIONS: Pleural Mesothelioma; Malignant Pleural Mesothelioma
Keywords: cisplatin; pleurectomy; decortication; heated cisplatin
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Cisplatin; sodium thiosulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Cisplatin — Given as a heated one-hour lavage to the hemithorax after surgery.
Drug: Sodium Thiosulfate — Given intravenously over 6 hours after the cisplatin lavage.

SUMMARY:
The purpose of this study it to determine the safety and maximally tolerated dose (MTD) of cisplatin administered in the operating room and put into the chest and abdomen for one hour. We are also looking at the effects of heating the chemotherapy to a temperature of 42 degrees celsius.

DETAILED DESCRIPTION:
* Patients will undergo surgery with pleurectomy/decortication which entails the removal of the inner and outer skin of the lung, including the pleura overlying the pericardium and diaphragm. Resection of the pericardium and diaphragm are occasionally necessary to debulk the tumor. This surgery is part of standard care for pleural mesothelioma.
* After surgery, a one hour lavage with heated cisplatin will be administered to the hemithorax (and abdominal regions if the diaphragm is no longer present). The lung itself is not removed, only the diseased portion of the lung and surrounding areas with tumor.
* Immediately following the one-hour lavage, a six hour infusion of sodium thiosulfate will begin to help reduce the side effects of the cisplatin.
* Patients will remain hospitalized until they have recovered from surgery (usually 7-14 days).
* Patients will return to the hospital three months after their surgery to have fluid drawn from their chest via an ultrasound guided thoracentesis. This is called a saline wash.
* Patients will be in the study actively for three months. This includes a 2-week and 4-week post-operative follow-up in which blood work is performed. As well as a 3-month follow-up for the saline wash. Long-term follow-up includes computed tomography of the chest and abdomen every 6 months to assess recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologic confirmation of malignant pleural mesothelioma
* Patients who are able to tolerate surgical cytoreduction but unable to undergo extrapleural pneumonectomy due to poor cardiopulmonary reserve or tumor invasion
* 18 years of age or older
* Malignancy is confined to the affected hemithorax.
* Grossly normal cardiac function with an EKG showing no cardiomyopathy or acute changes
* Evidence of adequate renal and hepatic function
* Karnofsky performance status of 70% or greater

Exclusion Criteria:

* Extended disease outside the ipsilateral hemithorax as determined radiologically and intraoperatively
* Distant metastases
* Non-malignant systemic disease
* Active concomitant malignancy
* Psychiatric or addictive disorders which would preclude obtaining informed consent
* Prior treatment within the last 2 months, other than surgical resection for their current malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 1999-08; Primary Completion 2002-04 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
To determine the maximally tolerated dose of intracavitary cisplatin in patients with malignant pleural mesothelioma, | 3 years

SECONDARY OUTCOMES:
To quantitate the safety of intraoperative intrathoracic/intraperitoneal hyperthermic cisplatin | 3 years
to study the pharmacokinetics of cisplatin administered in this way. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: David J. Sugarbaker, MD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts